CLINICAL TRIAL: NCT05693844
Title: Phase I/II Study of Pan-T Booster Co-expressing MSLN CAR T Cell Therapy in Advanced/Metastatic Solid Tumors
Brief Title: Pan-T Booster Co-expressing MSLN CAR T Cell Therapy in Advanced/Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: UTC Therapeutics Inc. (Industry)
Responsible Party: Principal Investigator, Han weidong, Director of Biotherapeutic Department, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHN-PLAGH-BT-077
Record Dates: First submitted 2022-12-27; First posted 2023-01-23 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Advanced or Metastatic Solid Tumors
MeSH Terms: interventions — Albumin-Bound Paclitaxel; Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pan-T booster co-expressing MSLN CAR T cell (Experimental): Before the infusion of pan-T booster co-expressing MSLN CAR T cells, all enrolled patients need to undergo conditioning chemotherapy consisting of albumin-bound paclitaxel, cyclophosphamide, and fludarabine.
  Interventions: Biological: Pan-T booster co-expressing MSLN CAR T cell; Drug: Albumin-bound paclitaxel; Drug: Cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Biological: Pan-T booster co-expressing MSLN CAR T cell — Starting Dose: 1×10^6 cells/kg
Drug: Albumin-bound paclitaxel — Administered intravenously at dose of 100-200mg/m2 on day -5
Drug: Cyclophosphamide — Administered intravenously at a total dose of 15-30mg/kg on day -3 and day -2
Drug: Fludarabine — Administered intravenously at dose of 30mg/m2/d on day -3 and day -2

SUMMARY:
In preclinical study, investigators have demonstrated that the newly developed pan-T booster (harbouring CD40 agonist and one T cell costimulator agonist) co-expressing MSLN CAR T cell possess more powerful antitumor activity than previously reported MSLN-CAR T cells. In this clinical trial, enrolled patients receive an initial dose of pan-T booster co-expressing MSLN CAR T cells at 1×10^6 cells/kg based on the basic principle of dose escalation design, in order to evaluate the safety, feasibility, pharmacokinetics/pharmacodynamics, and efficacy of pan-T booster co-expressing MSLN CAR T cell in vivo.

DETAILED DESCRIPTION:
In this study, investigators have developed a novel CAR T cell system targeting mesothelin (MSLN) antigen, termed as Pan-T booster (harbouring CD40 agonist and one T cell costimulator agonist) co-expressing MSLN CAR T cell. Preclinical study demonstrated that this novel pan-T booster co-expressing MSLN CAR T cell possess more powerful antitumor activity than previously reported MSLN-CAR T cells. In this clinical trial, enrolled patients receive an initial dose of pan-T booster co-expressing MSLN CAR T cells at 1×10^6 cells/kg based on the basic principle of dose escalation design, in order to evaluate the safety, feasibility, pharmacokinetics/pharmacodynamics, and efficacy of pan-T booster co-expressing MSLN CAR T cell in vivo. The level of CAR-T cell expansion and the duration of expansion are important determining factors for subsequent dose escalation infusions (3×10^6 cells/kg and 6×10^6 cells/kg). Repeated infusion, immune checkpoint inhibitor (such as anti-PD1/PD-L1) or local therapy (radiotherapy) are allowed when patients achieve clinical benefit and the level of CAR-T cell expansion declines to low level.

In the 3 patients receiving the first dose treatment, we observed high levels of expansion of both total T cells and CAR T cells in the PB after CAR T cell infusion (CAR T > 300 per microliter, total T cells reaching 10 times the number of CAR T cells), one patient experienced a grade 2 pulmonary toxicity and transient liver dysfunction during the CAR T cell expansion period (infusion 14 days later), transient marked enlargement of the spleen, and required to be treated with glucocorticoids and ruxolitinib to control T cell toxicity. Efficacy monitoring showed that some target lesion clearance or reduction could be achieved within 2-4 weeks after CAR T infusion. Based on these observations, it was concluded that low-dose CAR T infusion (CAR+T cells 1×10^6 cells/kg) could achieve the sufficient level of CAR T cell expansion, and the initially planned CAR T dose escalation was dispensable. Subsequent patients after May 10th, 2024, will all be treated using 1×10^6 cells/kg dose.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age from 18 to 75 years with estimated life expectancy >3 months.
* 2. Histopathological confirmed advanced or metastatic solid tumors failed to at least first-line treatment or initially diagnosed advanced/metastatic solid tumors that have no NCCN guideline recommended standard first-line therapy. Mesothelin antigen expression percentage >＝10%.
* 3. Have at least one measurable target lesion.
* 4. Fresh solid tumor samples or formalin-fixed paraffin embedded tumor archival samples within 6 months are necessary; Fresh tumor samples are preferred. Subjects are willing to accept tumor rebiopsy in the process of this study.
* 5. Previous treatment must be completed for more than 4 weeks prior to the enrollment of this study, and subjects have recovered to <= grade 1 toxicity.
* 6. Have an Eastern Cooperative Oncology Group performance status (ECOG) of 0 or 2 at the time of enrollment.
* 7. Have adequate organ function, which should be confirmed within 2 weeks prior to the first dose of study drugs.
* 8. Previous treatment with anti-PD-1/PD-L1 antibodies are allowed.
* 9. Ability to understand and sign a written informed consent document.
* 10. Women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, and up to 90 days after the last dose of the drug.

Exclusion Criteria:

* 1. Active, known or suspected autoimmune diseases.
* 2. Known brain metastases or active central nervous system (CNS). Subjects with CNS metastases who were treated with radiotherapy for at least 3 months prior to enrollment, have no central nervous symptoms and are off corticosteroids, are eligible for enrollment, but require a brain MRI screening.
* 3. Subjects are being treated with either corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of enrollment.
* 4. History of severe hypersensitive reactions to other monoclonal antibodies.
* 5. History of allergy or intolerance to study drug components.
* 6. Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results.
* 7. History or concurrent condition of interstitial lung disease of any grade or severely impaired pulmonary function.
* 8. Uncontrolled intercurrent illness, including ongoing or active systemic infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia (excluding insignificant sinus bradycardia and sinus tachycardia) or psychiatric illness/social situations and any other illness that would limit compliance with study requirements and jeopardize the safety of the patient.
* 9. History of human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS).
* 10. Pregnant or breast-feeding. Women of childbearing potential must have a pregnancy test performed within 7 days before the enrollment, and a negative result must be documented.
* 11. Previous or concurrent cancer within 3 years prior to treatment start EXCEPT for curatively treated cervical cancer in situ, non-melanoma skin cancer, superficial bladder tumors [Ta (non-invasive tumor), Tis (carcinoma in situ) and T1 (tumor invades lamina propria)].
* 12. Vaccination within 30 days of study enrollment.
* 13. Active bleeding or known hemorrhagic tendency.
* 14. Subjects with unhealed surgical wounds for more than 30 days.
* 15. Being participating any other trials or withdraw within 4 weeks.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-01-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment related adverse events | Up to 12 months since the initiation of MSLN targeted CAR T cell therapy
  Treatment related adverse events are defined as any medical events since the initiation of MSLN targeted CAR T cell therapy . CRS or CRES will be graded based on American Society for Transplantation and Cellular Therapy (ASTCT) criteria, and the others will be graded by CTCAE V5.0
Incidence of dose limiting toxicities (DLTs) | Up to 28 days since the initiation of MSLN targeted CAR T cell therapy
  Dose limiting toxicities are defined as MSLN targeted CAR T cell therapy related adverse events within the first 28 days that meet the following criteria: grade 3 or higher CRS or CRES, and any other grade 4 adverse events.

SECONDARY OUTCOMES:
Number and copy number of MSLN targeted CAR T cell | Up to 3 years
  Number and copy number of MSLN targeted CAR T cell are evaluated by number in peripheral blood and tumor tissue.
Objective response rate (ORR) | Up to 3 years
  Objective response rate includes complete response and partial response defined by investigators according to RECIST 1.1or iRECIST criteria.
Progression Free Survival (PFS) | Up to 3 years
  Progression Free Survival is defined as the time from the initiation of MSLN targeted CAR T cell therapy to documented disease progression or death.
Time to response (TTR) | Up to 3 years
  TTR is defined as the time from the initiation of MSLN targeted CAR T cell therapy to first assessed CR or PR by investigators according to RECIST 1.1or iRECIST criteria.
Duration of response (DOR) | Up to 3 years
  Duration of response is defined as the time from objective response until documented tumor progression among responders.
Overall Survival (OS) | Up to 3 years
  Overall Survival is defined as the time from the initiation of MSLN targeted CAR T cell therapy to documented disease progression or death.

CONTACTS AND LOCATIONS:
Overall Officials: Yangbin Zhao, PhD, Study Director — UTC Therapeutics Inc.
Locations (1):
- Kaichao Feng, Beijing, Beijing Municipality, China